CLINICAL TRIAL: NCT02815436
Title: The Effectiveness of Telephone Reminders and SMS Messages on Compliance With Colorectal Cancer Screening: An Open-label, Randomized Controlled Trial
Brief Title: Effectiveness of Tel and SMS Reminder on Compliance With CRC Screening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Martin Chi Sang Wong, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: Tel Compliance Study_Protocol
Record Dates: First submitted 2016-06-24; First posted 2016-06-28 (Estimated); Last update posted 2018-07-18 (Actual); Status verified 2018-07

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Telephone reminder (Active Comparator): subjects in this arm will receive a telephone reminder
  Interventions: Other: Telephone reminder
- SMS reminder (Active Comparator): Subjects in this arm will receive a SMS reminder
  Interventions: Other: SMS reminder
- No reminder (No Intervention): usual care, where no additional intervention will be offered

INTERVENTIONS:
Other: Telephone reminder — a personal, interactive telephone reminder by a centre colleague to remind return to the centre for taking faecal tubes for screening
  Arms: Telephone reminder
Other: SMS reminder — a one-way, SMS message sent from the centre to the screening participant's mobile phone
  Arms: SMS reminder

SUMMARY:
Colorectal cancer (CRC) is one of the major global health challenges. CRC is currently the third most common cancer in men and the second common in women worldwide, accounting for approximately 10% of all cancers.

Randomized controlled studies have shown that CRC screening using Faecal Occult Blood Testing (FOBT) is effective in reducing cancer mortality by 15-33%. Since yearly testing is recommended to maintain programmatic effectiveness, longitudinal adherence is a critical component of FOBT-based screening programs. The investigators previous study conducted in Hong Kong showed that the rate of compliance with CRC screening was declining since the first year of enrolment.

Nevertheless, it remains unknown whether interventions based on reminder systems could effectively enhance longitudinal compliance with FOBT, especially among those who have already enrolled in a CRC screening programme. Current evidence does not adequately compare whether interactive or one-way reminder messages are superior to usual care (i.e. no reminders).

DETAILED DESCRIPTION:
Colorectal cancer (CRC) is one of the major global health challenges. CRC is currently the third most common cancer in men and the second common in women worldwide, accounting for approximately 10% of all cancers. It leads to 8% of all cancer mortality in the world and it is the fourth most common cause of cancer deaths. There were 4,563 new cases and 3,893 new deaths in Hong Kong in 2012, while 47.4% of the new cases were diagnosed at stage III or above. In the past decades the Asia Pacific countries like China, South Korea, Japan, and Singapore have witnessed a two to three-fold rise in incidence, gradually catching up the figures in Western countries. The direct medical cost for the care of colorectal neoplasia was estimated US$45,115 for stage IV CRC in the initial year of care, bringing a substantial, global public health burden to the healthcare systems.

Randomized controlled studies have shown that CRC screening using Faecal Occult Blood Testing (FOBT) is effective in reducing cancer mortality by 15-33%. FOBT as a quick office-based procedure has the advantages of being non-invasive, inexpensive, acceptable, feasible, patient-friendly and devoid of needs for bowel preparation. A 25% relative risk reduction in CRC mortality was found for those attending at least one round of FOBT screening, according to a systematic review conducted in 2007. Guidelines from the US Preventive Services Task Force, the European Nations, the Asia Pacific Consensus statements and other authorities recommended FOBT as one of the first-line screening modalities, especially in resource-limited regions. Since yearly testing is recommended to maintain programmatic effectiveness, longitudinal adherence is a critical component of FOBT-based screening programs. The investigators previous study conducted in Hong Kong showed that the rate of compliance with CRC screening was declining since the first year of enrolment.

Nevertheless, it remains unknown whether interventions based on reminder systems could effectively enhance longitudinal compliance with FOBT, especially among those who have already enrolled in a CRC screening programme. Current evidence does not adequately compare whether interactive or one-way reminder messages are superior to usual care (i.e. no reminders).

ELIGIBILITY:
Inclusion Criteria:

* Subjects who joined the bowel cancer screening programme in the CUHK JC Bowel Cancer Education Centre who are expected to follow-up and return to the centre for annual Fecal Occult Blood Test.

Exclusion Criteria:

* Subjects who have medical conditions rendering them unable to understand telephone or SMS messages.
* Subjects without mobile phone

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2016-04; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Rate of completion of FOBT in the year of receiving the interventions/control | 1 year

SECONDARY OUTCOMES:
Rate of return of FOBT tubes in the year of receiving the interventions/control | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Martin Wong, MD, Principal Investigator — CUHK
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No